CLINICAL TRIAL: NCT05101200
Title: Dose Response of Neural Mobilization on Hamstring Flexibility in Patients With Non-specific Low Back Pain
Brief Title: Dose Response of Neural Mobilization on Hamstring Flexibility in Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rabia Liaquat
Record Dates: First submitted 2021-10-19; First posted 2021-11-01 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Non-specific Low Back Pain
Keywords: Neural Mobilization Technique; Oswestry Disability Index; Active Knee Extension Test; Numeric Pain Rating Scale; Lumbar flexion by Schober method

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Dose Neural Mobilization Technique (Experimental): Patients in this Group will receive High Dose Neural Mobilization Technique
  Interventions: Other: High Dose Neural Mobilization Technique
- Low Dose Neural Mobilization Technique (Experimental): Patients in this Group will receive Low Dose Neural Mobilization Technique
  Interventions: Other: Low Dose Neural Mobilization Technique

INTERVENTIONS:
Other: High Dose Neural Mobilization Technique — Patients in This Group will receive the high dose neural mobilization along with hot pack, strengthening exercises, Neural mobilization technique (slump, sciatic). Participants in the NMG will be asked to actively perform knee extension, ankle dorsiflexion, and head extension in a slumped posture (body and neck semi flexion) followed by simultaneous ankle plantar flexion together with knee and head flexion, Hot pack for 15 minutes, Strengthening exercises of muscles with 10 /8sets. Strengthening exercises of quadriceps with10 rep/8sets, Static stretching exercise for hamstring muscle with 10 rep/8sets, Group A will be given session of 40 min/day, 2 days/week for 4 weeks.
  Arms: High Dose Neural Mobilization Technique
Other: Low Dose Neural Mobilization Technique — Patients in this Group will receive the same treatment as group A but with less intensity and low dosage. Hot pack: 15 minutes, Strengthening exercises of muscles with 10 rep/4sets, Static stretching exercise for hamstring muscle with 10 rep/4sets. Group B will be given session of 40min/day, 2 days/week for 4weeks.
  Arms: Low Dose Neural Mobilization Technique

SUMMARY:
This study will be a randomized control trial and will be conducted in Riphah International Hospital, National orthopedic and specialist hospital, Riphah international hospital and Chambeli institute of physiotherapy. A sample of 34 participants will be taken. Participants will be randomized into Group A and Group B through lottery method. Group A will receive High Dose Neural Mobilization Technique, Hot pack for 15 minutes, strengthening exercises with 10rep/8sets , strengthening exercises for quadriceps and static stretching exercise for hamstring with 10 rep/8sets, While Group B will receive Low Dose Neural Mobilization Technique with minimal intensity, hot pack: 15 minutes, strengthening exercises with 10rep/4sets. Both groups will be given session of 40 min/day, 2 days/week for 4 weeks, assessment will be done at baseline, at the end of 1st week, 2nd week, 3rd week & at the end of 4th week. The outcome measure will be Numeric Pain Rating Scale (NPRS), Oswestry Disability Index (ODI), Active Knee Extension test (AKE) and Lumbar flexion by Schober method. Data will be analyzed be SPSS 22.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain > 3 months
* No exercises for last 6 months
* Non-specific LBP in its sub-acute & chronic phase

Exclusion Criteria:

* Specific causes of LBP (disc herniation, lumbar stenosis, spinal deformity, fracture, spondylolisthesis),
* Central or peripheral neurologic signs
* Systemic illness (tumor and rheumatologic diseases),
* Psychiatric and mental deficits.
* Patients who had undergone operations within 6 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 4 Weeks
  The Numeric Pain Rating Scale that is a uni-dimensional measure of pain intensity in adults. The 11-point numeric scale ranges from '0' representing one pain extreme (no pain) to '10' representing the other pain extreme (or "worst pain imaginable"). The intrarater reliability with ICC = 0.67.
Oswestry Disability Index (ODI) | 4 Weeks
  Oswestry Low Back Pain Disability Index(ODI) is a questionnaire reported by the patient itself for low back pain. The questionnaire into ten sections is divided and used to assess daily living activities limitations. Scored on scales of 0- 5 for each section, greatest disability is represented by 5. To calculate index summed scores is divided by the total score, then by 100 multiplied and as percentage it is expressed. With degree of disability associated are the scores indicating minimal to bed bound disability. 0% to 20% scores shows minimal disability, moderate disability indicated by scores from 20% to 40%, severe disability indicated by from 40% to 60% scores, 60% to 80% indicates crippled; and bedbound or exaggerating indicated by scores from 80% to 100%. Test-retest has high reliability (r = 0.83 to 0.99).
Active Knee Extension test for hamstring flexibility | 4 Weeks
  AKE test as known as active knee extension test is used to assess the flexibility and available Range of motion of hamstring muscle.The range of active knee extension in the position of hip flexion is easily assessed. M. Shamsi, Meriam et.al discussed the reliability and validity of this test and proved it as a valid tool for measurement of shortness in hamstring muscle.
Lumbar flexion by Schober method | 4 weeks
  For the measurement of OST, the participant stood erect while the lumbosacral junction was marked as indicated by the dimples of Venus. A second mark was placed 10 cm above the junction. The participant was then asked to bend forward as far as possible, and the stretched distance was indicated as the OST in cm.

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmed Awan, Ms-OMPT, Principal Investigator — Riphah International University
Locations (1):
- National orthopedic and specialist hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No